CLINICAL TRIAL: NCT01877057
Title: Assessment of the Effects of Gastric Degradation-protected Pea Protein Extract on Mucosal Satiety Hormone Release by Human Duodenal Tissue
Brief Title: Protected Pea Protein Extract and Satiety Hormone Release
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Bouke Salden, Medical Degree, Maastricht University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 133001
Record Dates: First submitted 2013-06-05; First posted 2013-06-13 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Obesity; Overweight
Keywords: Pea protein; Satiety hormone; Ussing Chamber
MeSH Terms: conditions — Obesity; Overweight | interventions — Saturn

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Saturn (Experimental): For the different prototypes of pea protein extract used in this study pea protein NUTRALYS F85M or F85G, Acacia Gum 381A or 396I and water will be used.
  Interventions: Dietary Supplement: Saturn

INTERVENTIONS:
Dietary Supplement: Saturn
  Other Names: Protected pea protein

SUMMARY:
The increasing prevalence of overweight and obesity among the population contributes to increased incidences of chronic metabolic diseases. Healthcare costs related to these diseases are rising; prevention or delay of onset of disorders associated with overweight is needed. Food ingestion exerts a transient suppressive effect on appetite and further food intake by releasing gastrointestinal hormones. Proteins have been shown to be more satiating than carbohydrates and fat. Intraduodenal administration (via a naso-duodenal intubation) of pea protein has been shown to reduce food intake and increase satiety hormone levels in humans, in contrast to orally dosed (unprotected) pea protein. In the present study we aim to investigate the effects of human gastric fluid on the degradability of five different protected pea protein products. Further, in an ex vivo experiment on freshly obtained human duodenum tissue applying Ussing chamber technology; we aim to investigate the intestinal satiety hormone release by the five different prototypes. The prototype that is less degraded by human gastric fluid and is most effective in intestinal satiety hormone release will be used in a future clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men/women
* BMI between 18 and 25 kg/m2
* Consistently stable body weight for at least 6 months (± 2 kg)

Exclusion Criteria:

* Type 2 diabetes mellitus (defined as fasting plasma glucose ≥ 7.0 mmol/L);
* Gastroenterological diseases or abdominal surgery (uncomplicated appendectomy, cholecystectomy and hysterectomy allowed, and other surgery upon judgment of the principle investigator);
* Cardiovascular diseases, cancer, liver or kidney malfunction, auto-immune diseases, disease with a life expectancy shorter than 5 years;
* Abuse of products; alcohol (>20 alcoholic consumptions per week) and drugs
* Smoking
* Plans to lose weight or following a hypocaloric diet;
* Use of any medication, including vitamin supplementation, except oral contraceptives, within 14 days prior to testing;
* Regular use of laxation products;
* Use of antibiotics in the 90 days prior to the start of study.
* Administration of investigational drugs or participation in any scientific intervention study which may interfere with this study (to be decided by the principle investigator), in the 90 days prior to the study
* Known pregnancy, lactation (checked by a pregnancy test before start of study)
* Blood donation within 3 months before study period
* Self-admitted HIV-positive state

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
To measure the release of satiety hormones (CCK, PYY, GLP-1) by intestinal mucosa in respons to five different protected pea protein extracts. | In Ussing Chamber at baseline
To measure the release of satiety hormones (CCK, PYY, GLP-1) by intestinal mucosa in respons to five different protected pea protein extracts. | In Ussing Chamber after 240 minutes

SECONDARY OUTCOMES:
To measure the degradability of the different prototypes by human gastric fluid, tested in an in vitro setting. | At baseline
  First, in vitro digestion will be conducted for the gastro-resistent protein in order to calculate the degree of hydrolysis of food proteins by o-phthaldialdehyde method (OPA). First, OPA solution and serine standard solution will be prepared. Samples are analyzed after the in vitro digestion. Measurements are made on 96 well microplates, each sample is analyzed twice. The absorbance is measured on spectrophotometer. The degree of hydrolysis corresponds to the amount of amino groups released during enzymatic digestion.

CONTACTS AND LOCATIONS:
Overall Officials: A.A.M. Masclee, Professor, Principal Investigator — Department of Internal Medicine, Division of Gastroenterology-Hepatology
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands